CLINICAL TRIAL: NCT04567342
Title: Effect of Varied Outreach Methods on Appointment Scheduling, Appointment Completion, and Receipt of MMR Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2020-0769
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Preventable Disease, Vaccine; Health Care Utilization
MeSH Terms: conditions — Vaccine-Preventable Diseases; Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Other: 1 automated message; Other: No personal contact attempt
- Arm 2 (Experimental)
  Interventions: Other: 2 automated messages; Other: No personal contact attempt
- Arm 3 (Experimental)
  Interventions: Other: 1 automated message; Other: 1 personal contact attempt
- Arm 4 (Experimental)
  Interventions: Other: 2 automated messages; Other: 1 personal contact attempt

INTERVENTIONS:
Other: 1 automated message — Parents of eligible patients will receive 1 HIPAA compliant automated call or text reminder (based on preference recorded in EHR) that their child is due for a checkup and information on how to schedule an appointment.
  Arms: Arm 1; Arm 3
Other: 2 automated messages — Parents of eligible patients will receive 2 HIPAA compliant automated call or text reminders (based on preference recorded in EHR) that their child is due for a checkup and information on how to schedule an appointment.
  Arms: Arm 2; Arm 4
Other: No personal contact attempt — No personal contact attempts will be made.
  Arms: Arm 1; Arm 2
Other: 1 personal contact attempt — Parents of eligible patients will receive a text from a medical assistant informing them that their child is due for a check up. This will be followed by personal call from the medical assistant to assist the parent with scheduling an appointment.
  Arms: Arm 3; Arm 4

SUMMARY:
Our objective is to determine the effectiveness of varied outreach methods (e.g. automated reminder calls/text messages with or without personalized calls/texts) to children age 12-14 months or 4 years old who are due for a WCC visit and don't have one scheduled in the next 45 days on the outcomes of appointment scheduling, appointment completion, and receipt of the MMR vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age: 12-14 months old OR 4 years old
* Has not yet received first MMR (for 12-14 month olds) OR second MMR (for 4 year olds)
* Has not had a well child check in past 365 days (for 4 year olds)
* No appointment scheduled in the next 45 days
* Parent preferred language = English or Spanish

Exclusion Criteria:

* Phone number not available in electronic medical record

Ages: 12 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1312 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B Brinkman, MD, Study Director — Cincinnati Children's
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Started | 329 | 328 | 328 | 327
Completed | 329 | 328 | 328 | 327
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Total
Number analyzed (Participants) | 329 | 328 | 328 | 327 | 1312
Age, Customized [Count of Participants; unit: Participants]
  12 m.o. | 64 | 62 | 61 | 60 | 247
  13 m.o. | 38 | 40 | 37 | 41 | 156
  14 m.o. | 15 | 15 | 18 | 15 | 63
  4 y.o. | 212 | 211 | 212 | 211 | 846
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 164 | 152 | 157 | 610
  Male | 192 | 164 | 176 | 170 | 702
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 16 | 23 | 58
  Not Hispanic or Latino | 313 | 315 | 309 | 296 | 1233
  Unknown or Not Reported | 7 | 3 | 3 | 8 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 2 | 4 | 1 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 3 | 3
  Black or African American | 241 | 252 | 248 | 232 | 973
  White | 54 | 45 | 47 | 53 | 199
  More than one race | 19 | 18 | 16 | 14 | 67
  Unknown or Not Reported | 13 | 9 | 16 | 21 | 59
Region of Enrollment [Number; unit: participants]
  United States | 329 | 328 | 328 | 327 | 1312

OUTCOME MEASURES:

1. Primary Outcome: Receipt of MMR Vaccination
Description: MMR administered to child (Yes or No) based on electronic health record documentation
Time Frame: By 15 months of age (for children who are 12-14 months old), or within 3 months of receiving intervention (for children age 4 years old)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 329 | 328 | 328 | 327
Participants | 92 | 77 | 99 | 104
Statistical Analysis 1: Comparison: Arm 1 vs Arm 3; Test type: Superiority; p = 0.531, Regression, Logistic; Risk Ratio (RR) = 1.08, 95% CI 2-sided [0.85 to 1.37]; Arm 3 vs. Arm 1
Statistical Analysis 2: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p = 0.189, Regression, Logistic; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.65 to 1.09]; Arm 2 vs. Arm 1
Statistical Analysis 3: Comparison: Arm 2 vs Arm 3; Test type: Superiority; p = 0.054, Regression, Logistic; Risk Ratio (RR) = 1.29, 95% CI 2-sided [0.10 to 1.66]; Arm 3 vs. Arm 2
Statistical Analysis 4: Comparison: Arm 3 vs Arm 4; Test type: Superiority; p = 0.654, Regression, Logistic; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.84 to 1.32]; Arm 4 vs. Arm 3
Statistical Analysis 5: Comparison: Arm 2 vs Arm 4; Test type: Superiority; p = 0.018, Regression, Logistic; Risk Ratio (RR) = 1.36, 95% CI 2-sided [1.05 to 1.74]; Arm 4 vs. Arm 2
Statistical Analysis 6: Comparison: Arm 1 vs Arm 4; Test type: Superiority; p = 0.283, Regression, Logistic; Risk Ratio (RR) = 1.14, 95% CI 2-sided [0.90 to 1.44]; Arm 4 vs. Arm 1

2. Secondary Outcome: Appointment Scheduled
Description: Appointment scheduled (Yes or No) based on electronic health record documentation
Time Frame: Within 2 weeks of receiving intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 329 | 328 | 328 | 327
Participants | 50 | 41 | 96 | 103
Statistical Analysis 1: Comparison: Arm 1 vs Arm 3; Test type: Superiority; p < 0.01, Regression, Logistic; Risk Ratio (RR) = 1.93, 95% CI 2-sided [1.42 to 2.62]; Arm 3 vs. Arm 1
Statistical Analysis 2: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p = 0.318, Regression, Logistic; Risk Ratio (RR) = 0.82, 95% CI 2-sided [0.56 to 1.21]; Arm 2 vs. Arm 1
Statistical Analysis 3: Comparison: Arm 2 vs Arm 3; Test type: Superiority; p < 0.01, Regression, Logistic; Risk Ratio (RR) = 2.34, 95% CI 2-sided [1.68 to 3.26]; Arm 3 vs. Arm 2
Statistical Analysis 4: Comparison: Arm 3 vs Arm 4; Test type: Superiority; p = 0.535, Regression, Logistic; Risk Ratio (RR) = 1.08, 95% CI 2-sided [0.85 to 1.36]; Arm 4 vs. Arm 3
Statistical Analysis 5: Comparison: Arm 2 vs Arm 4; Test type: Superiority; p < 0.01, Regression, Logistic; Risk Ratio (RR) = 2.52, 95% CI 2-sided [1.82 to 3.50]; Arm 4 vs Arm 2
Statistical Analysis 6: Comparison: Arm 1 vs Arm 4; Test type: Superiority; p < 0.01, Regression, Logistic; Risk Ratio (RR) = 2.07, 95% CI 2-sided [1.53 to 2.80]; Arm 4 vs. Arm 1

3. Secondary Outcome: Appointment Completed
Description: Appointment completed (Yes or No) based on electronic health record documentation
Time Frame: Within 8 weeks of receiving intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 329 | 328 | 328 | 327
Participants | 90 | 73 | 105 | 96
Statistical Analysis 1: Comparison: Arm 1 vs Arm 3; Test type: Superiority; p = 0.192, Regression, Logistic; Risk Ratio (RR) = 1.17, 95% CI 2-sided [0.92 to 1.48]; Arm 3 vs. Arm 1
Statistical Analysis 2: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p = 0.132, Regression, Logistic; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.62 to 1.06]; Arm 2 vs. Arm 1
Statistical Analysis 3: Comparison: Arm 2 vs Arm 3; Test type: Superiority; p < 0.01, Regression, Logistic; Risk Ratio (RR) = 1.44, 95% CI 2-sided [1.11 to 1.86]; Arm 3 vs. Arm 2
Statistical Analysis 4: Comparison: Arm 3 vs Arm 4; Test type: Superiority; p = 0.462, Regression, Logistic; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.73 to 1.16]; Arm 4 vs. Arm 3
Statistical Analysis 5: Comparison: Arm 2 vs Arm 4; Test type: Superiority; p = 0.039, Regression, Logistic; Risk Ratio (RR) = 1.32, 95% CI 2-sided [1.01 to 1.72]; Arm 4 vs. Arm 2
Statistical Analysis 6: Comparison: Arm 1 vs Arm 4; Test type: Superiority; p = 0.570, Regression, Logistic; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.84 to 1.37]; Arm 4 vs. Arm 1

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
All-Cause Mortality (participants affected / at risk) | 0/329 | 0/328 | 0/328 | 0/327
Serious Adverse Events (participants affected / at risk) | 0/329 | 0/328 | 0/328 | 0/327
Other Adverse Events (participants affected / at risk) | 0/329 | 0/328 | 0/328 | 0/327

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT04567342/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT04567342/SAP_001.pdf